CLINICAL TRIAL: NCT07342959
Title: Technique and Preliminary Results of Medial Epicondyle Fracture Fixation Using Anchors and Review of the Literature
Acronym: Epicondyle
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9814
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Medial Epicondyle Fractures of the Elbow
Keywords: Medial Epicondyle Fractures of the Elbow; Anchor Fixation; Fractures of the humerus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medial epicondyle fractures of the humerus account for 11 to 20% of elbow fractures in children and adolescents.

The therapeutic strategy remains controversial, ranging from conservative treatment to surgical fixation depending on the degree of displacement and joint instability.

Conventional surgical management of these fractures generally involves fixation with screws or pins. However, the occurrence of certain complications, such as hardware migration, soft tissue irritation, the risk of iatrogenic comminution of small bone fragments, and the need for implant removal, has led to the exploration of alternatives, including the use of anchor fixation.

This technique involves inserting an anchor with sutures into the bone to ensure stable fixation of the fragment, while reducing the risk of comminution and avoiding the need for subsequent removal of the material.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient (under 15 years of age)
* Admitted for recent displaced fractures of the medial epicondyle of the elbow
* Treated in the pediatric surgery department at Hautepierre Hospital
* Fractures requiring surgical treatment with anchor fixation.

Exclusion Criteria:

* Non-displaced fractures
* Open fractures and associated fractures

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient (under 15 years of age) admitted for recent displaced fractures of the medial epicondyle of the elbow
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score (MEPS) | Up to 12 months
  What the Mayo Performance Status (MEPS) measures:
  It assigns points (out of 100) based on:
  * Pain
  * Elbow mobility
  * Stability
  * Ability to perform everyday activities
  Interpretation of results:
  * 90-100 points: Excellent
  * 75-89 points: Good
  * 60-74 points: Average
  * <60 points: Poor

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Pédiatrique - CHU de Strasbourg - France, Strasbourg, France